CLINICAL TRIAL: NCT00778765
Title: Comparative, Randomized, Single-Dose, 2-Way Crossover Bioavailability Study of Ranbaxy and Parke-Davis (Neurontin®) 400 mg Gabapentin Capsules in Healthy Adult Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Gabapentin 400 mg Capsules Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA01820
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence gabapentin fed conditions
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 400 mg Gabapentin Capsules of Ranbaxy
  Interventions: Drug: 400 mg Gabapentin Capsules
- 2 (Active Comparator): Neurontin® 400 mg Gabapentin Capsules
  Interventions: Drug: 400 mg Gabapentin Capsules

INTERVENTIONS:
Drug: 400 mg Gabapentin Capsules

SUMMARY:
To compare the single-dose oral bioavailability of metformin HCI liquid 500 mg/5 mL of Ranbaxy with Glucophage® 1000 mg tablets of Bristol-Myers, USA following administration of a 1000 mg dose in healthy, adult, male and female volunteers under fasting conditions

DETAILED DESCRIPTION:
This was an open-label, randomized, single-dose, 2-way crossover, relative bioavailability study performed on 24 healthy adult volunteers and 2 alternates. All 26 subjects completed the clinical phase of the study. In each period, subjects were housed from the evening before dosing until after the 36-hour blood draw. Single oral 400 mg doses were separated by a washout period of 7 days A total of 24 healthy adult volunteers and 2 alternates (17 males and 9 non-pregnant females) enrolled in and completed the clinical phase of the study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers, 18-55 years of age
2. Weighing at least 52 kg for males and 45 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983)
3. Medically healthy subjects with clinically normal laboratory profiles
4. Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the study and throughout the study or be using one of the following acceptable birth control methods:

   * surgically sterile (bilateral tubal ligation, hysterectomy bilateral oophorectomy) 6 months minimum
   * IUD in place for at least 3 months
   * barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the start of the study and throughout the study
   * surgical sterilization of the partner (vasectomy for 6 months minimum)
   * hormonal contraceptives for at least 3 months prior to the start of the study

   Other birth control methods may be deemed acceptable. Postmenopausal women with amenorrhea for at least 2 years will be eligible.
5. Voluntarily consent to participate in the study.

Exclusion Criteria:

Subject candidates must not be enrolled in the study if they meet any of the following criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
2. In addition, history or presence of:

   * alcoholism or drug abuse within the past 2 years
   * hypersensitivity or idiosyncratic reaction to anticonvulsants
3. Female subjects who are pregnant or lactating
4. Subjects who have been on an abnormal diet (for whatever reason) during the 30 days prior to the first dose
5. Subjects who, through completion of the study, would have donated in excess of:

   * 500 mL of blood in 14 days, or
   * 500 - 750 mL of blood in 14 days (unless approved by the Principal Investigator)
   * 1000 mL of blood in 90 days
   * 1250 mL of blood in 12 days
   * 1500 mL of blood in 180 days
   * 2000 mL of blood in 270 days
   * 2500 mL of blood in I year
6. Subjects who have participated in another clinical trial within 28 days prior to the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-09; Primary Completion 2002-10 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Saint-Laurent, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html